CLINICAL TRIAL: NCT01168193
Title: Evaluation of Surgical Complications Using a Novel Grading System - A Prospective Single Arm Study
Brief Title: Evaluation of Surgical Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Hagai Mazeh, MD, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Complications-HMO-CTIL
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Post Operative Complications
Keywords: surgery; post operative; complications; length of stay

ARMS (1):
- Patients that underwent surgery (Other): Single arm
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Surgical complications may be very serious and are often under-reported. The aim of this study it to document and study all the postoperative complications at our department during one year using a novel grading system.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing surgery at our department.
* No gender difference.

Exclusion Criteria:

* Age - less than 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of complications | 1 year
  all post operative complications will be included

CONTACTS AND LOCATIONS:
Overall Officials: Haggi Mazeh, MD, Principal Investigator — Hadassah Medical Organization